CLINICAL TRIAL: NCT01379391
Title: A Phase IV, Open-label, Prospective, Multicenter Study of the Efficacy and Safety of Recombinant Human Thrombopoietin Injection (rHuTPO, TPIAO)on Platelet Engraftment in Allogeneic Hematopoietic Stem Cell Transplantation in China
Brief Title: Efficacy and Safety of rHuTPO on Platelet Engraftment After Allo-HSCT
Acronym: TPO
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Guangdong Provincial People's Hospital (Other); Guangdong No.2 Provincial People's Hospital (Other); Guangzhou General Hospital of Guangzhou Military Command (Other); Guangzhou Overseas Chinese Hospital,Guangdong (Unknown); Zhongshan People's Hospital, Guangdong, China (Other); Southern Medical University, China (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TPO-HSCT-2011
Record Dates: First submitted 2011-06-20; First posted 2011-06-23 (Estimated); Last update posted 2015-10-09 (Estimated); Status verified 2015-09

CONDITIONS: Allogeneic Hematopoietic Stem Cell Transplantation; Myeloablative; Delayed Platelet Engraftment
Keywords: Allogeneic Hematopoietic Stem Cell Transplantation; Platelet Engraftment; TPO
MeSH Terms: interventions — Thrombopoietin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TPO (Active Comparator): Patients received myeloablative Allo-HSCT with platelet lower than 20G/L on +14d post-transplantation. Patient enrolled in TPO arm will recieved Recombinant Human Thrombopoietin (rHTPO) treatment fro 14 days.
  Interventions: Drug: Recombinant Human Thrombopoietin (rHTPO)
- TPO-Free Arm (No Intervention): No TPO intervention

INTERVENTIONS:
Drug: Recombinant Human Thrombopoietin (rHTPO) — Patients received allogeneic myeloablative hematopoietic stem cell transplantation with platelet count lower than 20G/L on +14 days after Allo-HSCT, met the above enrollment criteria and signed the informed consent forms are eligible subjects.
  Administration method of rHuTPO: 300U/kg/d by percutaneous injection; Timing: d14 to d28 after Allo-HSCT.
  Arms: TPO

SUMMARY:
Factors influencing platelet engraftment after allogeneic hematopoietic stem cell transplantation (Allo-HSCT) includes previous chemotherapy courses, conditioning regimen, HLA compatibility, source of stem cell, CD34+ cell count, infection of virus/bacteria/fungal, graft-versus-host disease (GVHD), etc. Large-scaled clinical trials have demonstrated that platelet count below 20G/L on 14 days after transplantation is an predictive factor for delayed platelet engraftment, which lead to increased platelet infusion requirement and high risk of bleeding. Multivariable survival analysis indicated that delayed platelet engraftment in Allo-HSCT is independent predictive factor for transplantation related mortality (TRM). But effective treatment approaches for delayed platelet recovery after Allo-HSCT are still lacking now.

Recombinant human thrombopoietin (rHuTPO) is a fully modified recombinant human thrombopoietin accurately expressed in mammalian cells. The rHuTPO agent manufactured by the 3Bio Pharmaceutical Limited Liability Company (LLC) in Shenyang is approved by the State Food and Drug Administration (SFDA) of China in 2005 and is the first rHuTPO agent available globally. RHuTPO was approved for for immune thrombocytopenia and chemotherapy-related thrombocytopenia in China. Animal experiments showed that TPO-mobilizing stem cell could promote platelet engraftment in Allo-HSCT in mice. As for efficacy and safety of TPO on platelet engraftment after Allo-HSCT, it's marginally addressed in clinical trials.

Based on preliminary research results, investigator designed a phase IV, open-label, prospective, multicenter Study of the efficacy and safety of recombinant human thrombopoietin injection (rHuTPO, TPIAO)on platelet engraftment in Allo-HSCT in China.

ELIGIBILITY:
Inclusion Criteria:

1. Ages: 18 years to 65 years.
2. Patients received myeloablative allogeneic hematopoietic stem cell transplantation from related or non-related, HLA compatible or incompatible donors. History controls or concurrent controls are used.
3. The platelet count is lower than 20G/L on +14d post-transplant .
4. The informed consent form has been signed.
5. The following exclusion criteria are excluded.

Exclusion Criteria:

1. Patients received non-myeloablative hematopoietic stem cell transplantation.
2. Patients with severe cardio-cerebral diseases with over grade III A YHA cardiac function or with past history of coronary heart disease, cerebral thrombosis, cerebral arteriosclerosis, etc.
3. Patients with severe hepatic or renal dysfunction with more than 5 times the upper limit of normal range (ULN) of serum ALT or AST levels, or with more than 5 times the upper limit of normal range (ULN) of serum TBIL level or less than 40% of normal prothrombin time activity (PTA); or with more than 3 times the ULN of serum Cr.
4. Patients with history of deep vein thrombosis within 8 weeks of enrollment.
5. Patients with hepatic obstructive venous disease without recovery within 2 weeks of enrollment.
6. Patients with thrombotic microangiopathy without recovery within 2 weeks of enrollment.
7. Patients with capillary leaking syndrome without recovery within 2 weeks of enrollment.
8. Patients with other conditions considered unsuitable for the study.
9. Patients with hypercoagulopathy condition with two or more of these criteria: INR lower than 0.82, APTT lower than the lower limit of normal values (23 seconds) or PT lower than the lower limit of normal values (10 seconds).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2010-06; Primary Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Total Response Rate to TPO | 4 weeks
  Response Rate is selected as primary outcome for measuring efficacy of TPO for patients with delayed platelet engraftment after Allo-HSCT.
  Markedly response: Platelet count of more than 50G/L in complete blood count on +28d post-transplantation after finishing 14-day course of TPO intervention, or PLT≥100G/L within the 14-day course.
  Response: PLT 20-50G/L on +28 day after completing the 14-day course. No response: PLT <20G/L on +28 day after completing the 14-day course.

SECONDARY OUTCOMES:
Transplantation Related Mortality (TRM) | 1 year
  Transplantation related mortality (TRM) in two arms after Allo-HSCT.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Sun, MD, Principal Investigator — Department of Hematology, Nanfang Hospital
Locations (9):
- China (9):
  - Guangzhou General Hospital of Guangzhou Military Command, Guangzhou, Guangdong
  - Guangdong General Hospital, Guangzhou, Guangdong
  - First Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Guangdong No.2 Provincial People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital, Guangzhou, Guangdong
  - Guangzhou Overseas Chinese Hospital,Guangdong, Guangzhou, Guangdong
  - Third Affiliated Hospital, Sun Yat-Sen University, Guangzhou, Guangdong
  - Zhongshan People Hospital,Guangdong, Zhongshan, Guangdong

REFERENCES:
- See also: Website of Nanfang Hospital, Southern Medical University, Guangzhou, 510515, China. — http://www.nfyy.com